CLINICAL TRIAL: NCT05888103
Title: A 6 Month Randomized, Double-blind, Placebo-controlled Study Followed by a 6 Month Open- Label Extension to Assess the Efficacy and Safety of Inclisiran as Monotherapy in Chinese Adults With Low or Moderate ASCVD Risk and Elevated Low-density Lipoprotein Cholesterol
Brief Title: Efficacy and Safety of Inclisiran as Monotherapy in Chinese Adults With Low or Moderate ASCVD Risk and Elevated Low-density Lipoprotein Cholesterol.
Acronym: V-Mono China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CKJX839D12305
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Primary Hypercholesterolemia or Mixed Dyslipidemia
Keywords: Inclisiran; LDL-C; monotherapy; atherosclerotic cardiovascular disease; atheroma; Atherosclerosis; lipid; lipid lowering therapy (LLT); cholesterol; hypercholesteremia; mixed dyslipidemia; TC (total cholesterol); Apo B; non HDL-C; Lp(a); PCSK9; PCSK9 inhibitor; siRNA; low ASCVD risk; moderate ASCVD risk
MeSH Terms: conditions — Atherosclerosis; Plaque, Atherosclerotic; Hypercholesterolemia | interventions — ALN-PCS

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-blind, placebo-controlled, parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor Personnel participating in the study conduct were also blinded during the during core part of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inclisiran - Inclisiran (Experimental): Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) s.c administered on Day 1, Day 90, and Day 270, and placebo on Day 180
  Interventions: Drug: Inclisiran; Drug: Matching Placebo for Inclisiran
- Placebo- Inclisiran (Placebo Comparator): Placebo on Day 1 and Day 90 and Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) s.c on Day 180 and 270
  Interventions: Drug: Inclisiran; Drug: Matching Placebo for Inclisiran

INTERVENTIONS:
Drug: Inclisiran — Inclisiran s.c
  Other Names: KJX839
Drug: Matching Placebo for Inclisiran — Matching s.c. placebo
  Other Names: Placebo s.c.

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of inclisiran as a monotherapy in Chinese adults with low or moderate atherosclerotic cardiovascular disease (ASCVD) risk and elevated low-density lipoprotein cholesterol (LDL-C) who were not on any lipid lowering therapy.

DETAILED DESCRIPTION:
This study was designed as a randomized, double-blind, multi-center Phase III trial, with a placebo-controlled treatment period and an open label treatment period, to evaluate the efficacy and safety of inclisiran sodium 300 mg s.c. in participants aged 18 to 75 years with a low or moderate ASCVD risk and fasting LDL-C value of ≥ 130 mg/dL but < 190 mg/dL who were not on any lipid lowering therapy.

The study consisted of 3 parts:

* Screening: the screening period was up to 14 days to allow adequate time for the eligibility evaluations.
* Core Part: a double-blind, placebo-controlled treatment period of 180 days in which eligible participants were randomized 1:1 to receive either inclisiran sodium 300 mg s.c.

(inclisiran group) or matching placebo s.c. (control group) on Day 1 and Day 90. The end of core part (EOC) visit was conducted on Day 180. The database lock for the core part was planned to occur after all randomized participants have completed the EOC visit (or have discontinued from the study before EOC). The primary analysis was conducted after the database lock for the core part.

• Extension Part: an extended treatment period of 180 days. In the extension part, participants originally randomized to inclisiran in the core part were to continue the inclisiran treatment while participants initially randomized to placebo were to transit to the inclisiran. The extension part was to start from the Day 180 treatment dose (placebo in the inclisiran group and inclisiran for participants originally randomized to the control group).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Fasting LDL-C of ≥ 130 mg/dL but < 190 mg/dL
* Triglycerides ≤ 400 mg/dL
* Categorized as low or moderate ASCVD risk by the 2016 Chinese Guideline

Exclusion Criteria:

* Use of any LLT within 90 days prior to screening visit
* History of ASCVD
* Diabetes mellitus or fasting plasma glucose of ≥ 7.0 mmol/L or HbA1c ≥ 6.5%
* Secondary hypercholesterolemia, e.g. hypothyroidism or nephrotic syndrome

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- China (20):
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Zhongshan, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Hohhot, Inner Mongolia
  - Novartis Investigative Site, Changzhou, Jiangsu
  - Novartis Investigative Site, Xuzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Jinzhou, Liaoning
  - Novartis Investigative Site, Linyi, Shandong
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient level data and supporting clinical documents from eligible studies. these requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2932

RESULTS

PARTICIPANT FLOW:
Groups:
- Inclisiran - Inclisiran: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) s.c administered on Days 1, 90, and 270, and with matching placebo s.c administered on Day 180
- Placebo- Inclisiran: Placebo s.c administered on Days 1 and 90 and Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) s.c administered on Days 180 and 270
Period: Overall Study
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Started | 103 | 104
Completed extension part study | 98 | 101
Completed (Completed core part study) | 100 | 101
Not Completed | 3 | 3
Not completed — Participant decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran | Total
Number analyzed (Participants) | 103 | 104 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (9.97) | 47.7 (10.63) | 47.9 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 63 | 121
  Male | 45 | 41 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 103 | 104 | 207
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Low-density Lipoprotein Cholesterol (LDL-C) (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: Low-density lipoprotein cholesterol is a type of lipoprotein in the blood. Lipoproteins are particles made of lipids(fats) and proteins that carry fats through the bloodstream. Because of their structure, fats can't move through the blood on their own. So, lipoproteins carry fats to various cells in the body.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in LDL-C
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in LDL-C | -45.87 [-49.33 to -42.42] | 1.62 [-1.77 to 5.02]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -47.50, 95% CI 2-sided [-52.35 to -42.65]

2. Secondary Outcome: Absolute Change in LDL-C (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: as for outcome 1
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
mg/dL | -69.05 [-73.95 to -64.15] | 0.68 [-4.13 to 5.49]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -69.73, 95% CI 2-sided [-76.60 to -62.86]

3. Secondary Outcome: Percentage Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) (ng/mL) From Baseline at Day 150 - Core Analysis: Core Part
Description: Inclisiran is a double-stranded small interfering ribonucleic acid (siRNA) that causes degradation of protein convertase subtilisin/kexin type 9 (PCSK9) messenger RNA (mRNA) leading to the reduction of PCSK9 protein. The percentage change from baseline in PCSK9 at Day 150 was assessed.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in PCSK9
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in PCSK9 | -71.95 [-77.68 to -66.22] | 5.88 [0.24 to 11.52]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -77.83, 95% CI 2-sided [-85.86 to -69.80]

4. Secondary Outcome: Absolute Change in PCSK9 (ng/mL) From Baseline at Day 150 - Core Analysis: Core Part
Description: Inclisiran is a double-stranded small interfering ribonucleic acid (siRNA) that causes degradation of protein convertase subtilisin/kexin type 9 (PCSK9) messenger RNA (mRNA) leading to the reduction of PCSK9 protein.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
ng/mL | -217.14 [-230.15 to -204.13] | 9.47 [-3.24 to 22.17]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -226.61, 95% CI 2-sided [-244.77 to -208.45]

5. Secondary Outcome: Percentage Change in Total Cholesterol (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: Total cholesterol is a measure of all the cholesterol in the blood. It includes low-density lipoprotein (LDL), high-density lipoprotein (HDL) and a portion of triglycerides.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in total cholesterol
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in total cholesterol | -29.88 [-32.32 to -27.43] | 1.61 [-0.78 to 4.01]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -31.49, 95% CI 2-sided [-34.91 to -28.07]

6. Secondary Outcome: Absolute Change in Total Cholesterol (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: as for outcome 5
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
mg/dL | -68.82 [-74.37 to -63.28] | 2.64 [-2.80 to 8.09]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -71.46, 95% CI 2-sided [-79.24 to -63.69]

7. Secondary Outcome: Percentage Change in High-density Lipoprotein Cholesterol (HDL-C) (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: HDL-C stands for high-density lipoprotein cholesterol, often referred to as the "good" cholesterol. This is because HDL cholesterol helps remove other forms of cholesterol from the bloodstream. It picks up excess cholesterol in the blood and carries it back to the liver, where it is broken down and flushed out of the body.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in HDL-C
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in HDL-C | 12.24 [7.62 to 16.86] | 9.30 [4.74 to 13.86]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p = 0.3743, ANCOVA; LS Mean Difference = 2.94, 95% CI 2-sided [-3.55 to 9.42]

8. Secondary Outcome: Absolute Change in HDL-C (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: as for outcome 7
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
mg/dL | 4.66 [2.80 to 6.52] | 3.60 [1.76 to 5.43]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p = 0.4228, ANCOVA; LS Mean Difference = 1.07, 95% CI 2-sided [-1.54 to 3.68]

9. Secondary Outcome: Percentage Change in Non-HDL-C (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: Non-HDL cholesterol is a measure of all the "bad" types of cholesterol in the blood, excluding HDL cholesterol. It is calculated by subtracting HDL cholesterol from total cholesterol. Non-HDL cholesterol includes all the types of cholesterol other than HDL cholesterol, and higher levels of non-HDL cholesterol can increase the risk of cardiovascular disease.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in non-HDL-C
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in non-HDL-C | -40.71 [-43.57 to -37.85] | -0.14 [-2.93 to 2.66]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -40.57, 95% CI 2-sided [-44.57 to -36.57]

10. Secondary Outcome: Absolute Change in Non-HDL-C (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: as for outcome 9
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
mg/dL | -73.48 [-78.63 to -68.33] | -1.14 [-6.19 to 3.91]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -72.34, 95% CI 2-sided [-79.56 to -65.13]

11. Secondary Outcome: Percentage Change in Apolipoprotein B (ApoB) (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: Apolipoprotein B (ApoB) is a protein that helps carry fat and cholesterol through the body. It is encoded by the APOB gene. ApoB attaches to negative types of cholesterol that cause plaque buildup in blood vessels, which can lead to damage and heart disease.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in apolipoprotein B
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in apolipoprotein B | -36.63 [-39.40 to -33.86] | 0.21 [-2.50 to 2.93]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -36.84, 95% CI 2-sided [-40.72 to -32.96]

12. Secondary Outcome: Absolute Change in ApoB (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: as for outcome 11
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
mg/dL | -42.64 [-45.78 to -39.49] | -0.76 [-3.85 to 2.32]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -41.87, 95% CI 2-sided [-46.28 to -37.47]

13. Secondary Outcome: Percentage Change in Apolipoprotein A-1 (ApoA-1) (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: Apolipoprotein A1 (ApoA1) is the primary protein associated with high-density lipoprotein (HDL) particles, and plays a central role in reverse cholesterol transport. HDL cholesterol (HDL-C) and ApoA1 concentrations are inversely related to the risk for coronary artery disease (CAD).
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in apolipoprotein A-1
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in apolipoprotein A-1 | 5.11 [2.34 to 7.88] | 3.06 [0.33 to 5.79]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p = 0.3011, ANCOVA; LS Mean Difference = 2.05, 95% CI 2-sided [-1.84 to 5.93]

14. Secondary Outcome: Absolute Change in ApoA-1 (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: as for outcome 13
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
mg/dL | 6.44 [2.72 to 10.16] | 3.31 [-0.35 to 6.98]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p = 0.2403, ANCOVA; LS Mean Difference = 3.13, 95% CI 2-sided [-2.09 to 8.35]

15. Secondary Outcome: Percentage Change in Lipoprotein (a) (Lp(a)) (Nmol/L) From Baseline at Day 150 - Core Analysis: Core Part
Description: Often referred to as Lp(a), lipoprotein (a) is a type of lipoprotein that is genetically inherited and in high levels is a common independent risk factor for heart disease.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in lipoprotein (a)
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in lipoprotein (a) | -23.84 [-31.20 to -16.48] | 6.43 [-0.77 to 13.62]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -30.27, 95% CI 2-sided [-40.58 to -19.95]

16. Secondary Outcome: Absolute Change in Log-transformed Lp(a) (Nmol/L) From Baseline at Day 150 - Core Analysis: Core Part
Description: as for outcome 15
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
nmol/L | 0.68 [0.63 to 0.74] | 1.01 [0.93 to 1.09]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = 0.68, 95% CI 2-sided [0.60 to 0.76]

17. Secondary Outcome: Percentage Change in Triglyceride (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: Triglycerides are fats from the food we eat. Most of the fats we eat (like butter) are in triglyceride form. Extra calories, alcohol and sugar in the body turn into triglycerides. The body stores them in fat cells throughout the body.
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in Triglyceride
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
% change in Triglyceride | 3.49 [-4.44 to 11.43] | 0.48 [-7.01 to 7.97]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p = 0.5877, ANCOVA; LS Mean Difference = 3.01, 95% CI 2-sided [-7.88 to 13.91]

18. Secondary Outcome: Absolute Change in Triglyceride (mg/dL) From Baseline at Day 150 - Core Analysis: Core Part
Description: as for outcome 17
Time Frame: Baseline, Day 150
Population: Full analysis set - all treated participants
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
mg/dL | -15.32 [-31.86 to 1.22] | -7.36 [-23.67 to 8.94]
Statistical Analysis 1: Comparison: Inclisiran - Inclisiran vs Placebo- Inclisiran; Test type: Superiority; p = 0.5019, ANCOVA; LS Mean Difference = -7.96, 95% CI 2-sided [-31.17 to 15.26]

19. Secondary Outcome: Percentage Change in LDL-C (mg/dL) From Baseline at Day 330 - Final Analysis: Core Part + Extension Part
Description: as for outcome 1
Time Frame: Baseline, Day 330
Population: Full analysis set - all treated participants in the Inclisiran - Inclisiran group
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in LDL-C
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 0
% change in LDL-C | -45.45 [-48.57 to -42.34] |

20. Secondary Outcome: Absolute Change in LDL-C (mg/dL) From Baseline at Day 330 - Final Analysis: Core Part + Extension Part
Description: as for outcome 1
Time Frame: Baseline, Day 330
Population: Full analysis set - all treated participants in the Inclisiran - Inclisiran group
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 0
mg/dL | -67.55 [-72.39 to -62.72] |

21. Secondary Outcome: Number of Participants With Adverse Events (AEs) During Core Part
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject
Time Frame: Core part, from treatment start (Day 1) to Day 150
Population: Safety set - all treated participants in the core part
Measure: Count of Participants; unit: Participants
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
Participants
  Adverse events (AEs) | 73 | 70
  -Adverse events Treatment-related | 14 | 4
  Serious adverse events (SAEs) | 5 | 3
  -SAEs Treatment-related | 0 | 0
  Fatal SAEs | 0 | 0
  -Fatal SAEs Treatment-related | 0 | 0
  AEs leading to treatment discontinuation | 0 | 0
  -Treatment-related | 0 | 0
  AEs requiring additional therapy | 52 | 50

22. Secondary Outcome: Number of Participants With Adverse Events (AEs) During Extension Part
Description: as for outcome 21
Time Frame: Extension part, from Day 181, up to Day 360
Population: Final analysis - all treated participants in the extension part
Measure: Count of Participants; unit: Participants
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 100 | 101
Participants
  Adverse events (AEs) | 52 | 47
  -Adverse events Treatment-related | 9 | 15
  Serious adverse events (SAEs) | 1 | 2
  -SAEs Treatment-related | 0 | 0
  Fatal SAEs | 0 | 0
  -Fatal SAEs Treatment-related | 0 | 0
  AEs leading to treatment discontinuation | 0 | 0
  -Treatment-related | 0 | 0
  AEs requiring additional therapy | 36 | 28

23. Secondary Outcome: Number of Participants With Adverse Events (AEs) - Cumulative Data (Core + Extension Part)
Description: as for outcome 21
Time Frame: AEs are reported from first dose of study treatment until end of study treatment plus 30 days after the last study visit (or 90 days after the last administration of study drug, whichever is longer) up to a maximum timeframe of approximately 360 days
Population: Final analysis - all treated participants (Core + Extension part)
Measure: Count of Participants; unit: Participants
Arm/Group | Inclisiran - Inclisiran | Placebo- Inclisiran
Number analyzed (Participants) | 103 | 104
Participants
  Adverse events | 85 | 81
  -Adverse events Treatment-related | 18 | 18
  SAEs | 6 | 5
  -SAEs Treatment-related | 0 | 0
  Fatal SAEs | 0 | 0
  -Fatal SAEs Treatment-related | 0 | 0
  AEs leading to treatment discontinuation | 0 | 0
  -Treatment-related | 0 | 0
  AEs requiring additional therapy | 65 | 63

ADVERSE EVENTS:
Time Frame: AEs are reported from first dose of study treatment until end of study treatment plus 30 days after the last study visit (or 90 days after the last administration of study drug, whichever is longer) up to a maximum timeframe of approximately 360 days
Groups:
- Inclisiran - Inclisiran: Core Part: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran): core part
- Placebo - Inclisiran: Core Part: Placebo - inclisiran: core part
- Inclisiran - Inclisiran: Extension Part: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran): extension part
- Placebo - Inclisiran: Extension Part: Placebo - inclisiran: extension part
Arm/Group | Inclisiran - Inclisiran: Core Part | Placebo - Inclisiran: Core Part | Inclisiran - Inclisiran: Extension Part | Placebo - Inclisiran: Extension Part
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/104 | 0/100 | 0/101
Serious Adverse Events (participants affected / at risk) | 5/103 | 3/104 | 1/100 | 2/101
Other Adverse Events (participants affected / at risk) | 40/103 | 27/104 | 25/100 | 20/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran - Inclisiran: Core Part (N=103) | Placebo - Inclisiran: Core Part (N=104) | Inclisiran - Inclisiran: Extension Part (N=100) | Placebo - Inclisiran: Extension Part (N=101)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran - Inclisiran: Core Part (N=103) | Placebo - Inclisiran: Core Part (N=104) | Inclisiran - Inclisiran: Extension Part (N=100) | Placebo - Inclisiran: Extension Part (N=101)
Upper respiratory tract infection (Infections and infestations) | 25 | 17 | 14 | 9
Alanine aminotransferase increased (Investigations) | 6 | 3 | 5 | 4
Blood creatine phosphokinase increased (Investigations) | 7 | 6 | 6 | 7
Blood glucose increased (Investigations) | 10 | 7 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT05888103/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT05888103/SAP_001.pdf